CLINICAL TRIAL: NCT00094744
Title: A Randomized Trial Comparing Part-time Versus Full-time Patching for Severe Amblyopia
Brief Title: Trial Comparing Part-time Versus Full-time Patching for Severe Amblyopia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Roy W. Beck, M.D., Ph.D., Jaeb Center for Health Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-88; 2U10EY011751 (NIH)
Record Dates: First submitted 2004-10-22; First posted 2004-10-25 (Estimated); Last update posted 2010-09-09 (Estimated); Status verified 2010-09

CONDITIONS: Amblyopia
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 6hrs daily patching (Active Comparator): 6 hours per day of patching in the sound eye
  Interventions: Device: Eye patch
- Full-time daily patching (Active Comparator): Patching of the sound eye all but one waking hour
  Interventions: Device: Eye patch

INTERVENTIONS:
Device: Eye patch — adhesive eye patch used to cover the sound eye
  Other Names: Coverlet; Opticlude

SUMMARY:
The goals of this study are:

* To determine whether the visual acuity improvement obtained with part-time (6 hours) patching is equivalent to the visual acuity improvement obtained with full-time patching (all or all but one waking hour) for severe amblyopia.
* To develop more precise estimates than currently available for the visual acuity improvement that occurs during treatment of amblyopia with patching.
* To identify factors that may be associated with successful treatment of amblyopia with patching.

DETAILED DESCRIPTION:
Amblyopia is the most common cause of monocular visual impairment in both children and young and middle-aged adults. Patching has been the mainstay of amblyopia therapy. It is generally held that the response to treatment is best when it is instituted at an early age, particularly by age two or three, and is poor when attempted after eight years of age.

For severe amblyopia, it is generally accepted that occlusion with patching is the standard of care. Other modalities of treatment, such as atropine penalization and optical penalization, are widely considered insufficient as initial treatments for severe amblyopia. However, controversy exists with regard to how many hours per day of patching should be prescribed. Advocates of full-time patching purport that such a regimen is needed to restore visual acuity more rapidly and more effectively. Advocates of part-time patching believe it to be better tolerated by the child and family, therefore producing less stress on the parent-child relationship and producing better results through better compliance. Part-time patching may also promote the development of binocularity in patients who have "straight-eyes", reduce the chance of a straight-eyed patient developing manifest strabismus or losing stereopsis, and reduce the incidence of reverse- or occlusion-amblyopia.

The study is a randomized trial comparing daily patching regimes for children with severe amblyopia. It will consist of about 160 children. Patients in the severe (20/100 to 20/400) group will patch part-time (6 hours) or full-time (all or all but one waking hour) of each day for the 4 month study period. There are at least two follow up visits during the 4-month period. Visual acuity is the major study outcome. It is assessed at the 4-month exam.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be less than 7 years of age with the original cause of amblyopia as strabismus or anisometropia (a refractive error difference of more than one diopter between the two eyes.)
* Visual acuity in the amblyopic eye must be between 20/100 and 20/400.
* Visual acuity in the sound eye of 20/40 or better.
* There must be at least 3 lines of acuity difference between the two eyes.

Exclusion Criteria:

* Patching treatment (other than spectacles) within six months prior to enrollment and other amblyopia treatment of any type used within one month prior to enrollment.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2001-05; Primary Completion 2003-07 (Actual); Study Completion 2003-09 (Actual)

PRIMARY OUTCOMES:
Visual acuity improvement at 17wks. | 17 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael X Repka, M.D., Study Chair — Wilmer Eye Institute
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States

REFERENCES:
- [Background] Holmes JM, Kraker RT, Beck RW, Birch EE, Cotter SA, Everett DF, Hertle RW, Quinn GE, Repka MX, Scheiman MM, Wallace DK; Pediatric Eye Disease Investigator Group. A randomized trial of prescribed patching regimens for treatment of severe amblyopia in children. Ophthalmology. 2003 Nov;110(11):2075-87. doi: 10.1016/j.ophtha.2003.08.001. PMID 14597512
- [Derived] Repka M, Simons K, Kraker R; Pediatric Eye Disease Investigator Group. Laterality of amblyopia. Am J Ophthalmol. 2010 Aug;150(2):270-4. doi: 10.1016/j.ajo.2010.01.040. Epub 2010 May 8. PMID 20451898